CLINICAL TRIAL: NCT05544045
Title: Endovascular Treatment of Patients in China With the Surpass Streamline Flow Diverter for Unruptured Large and Giant Saccular Wide-Neck or Fusiform Intracranial Aneurysms in the Internal Carotid Artery
Brief Title: China Surpass Streamline Post-Market Study
Status: Terminated | Type: Observational
Why Stopped: Slow Enrollment
Sponsor: Stryker Neurovascular (Industry)
Collaborators: Stryker (Beijing) Healthcare Products Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: NV00050330
Record Dates: First submitted 2022-06-17; First posted 2022-09-16 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Aneurysm, Intracranial
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Surpass Streamline Flow Diverter System — The Surpass Streamline FDS is indicated for use in the endovascular treatment of adults (age 18 years or older) with unruptured large (≥ 10 mm) saccular, wide-neck (neck width ≥ 4 mm or dome/neck ratio < 2 mm) or fusiform intracranial aneurysms in the internal carotid artery from the petrous segment to the terminus arising from a parent vessel with a diameter ≥ 2.5 mm to ≤ 5.3 mm.

SUMMARY:
A multi-center, prospective, single-arm, non-randomized, post-market, observational study.

The primary objective of this study is to evaluate the long-term safety and efficacy of the Surpass Streamline Flow Diverter System (FDS) in the treatment of unruptured large and giant (≥ 10 mm) saccular wide-neck (neck width ≥ 4 mm) or fusiform intracranial aneurysms in the internal carotid artery from the petrous segment to the terminus arising from a parent vessel with a diameter ≥ 2.5 mm to ≤ 5.3 mm.

DETAILED DESCRIPTION:
The Surpass Streamline FDS is indicated for use in the endovascular treatment of adults (age 18 years or older) with unruptured large (≥ 10 mm) saccular, wide-neck (neck width ≥ 4 mm or dome/neck ratio < 2 mm) or fusiform intracranial aneurysms in the internal carotid artery from the petrous segment to the terminus arising from a parent vessel with a diameter ≥ 2.5 mm to ≤ 5.3 mm.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age ≥ 18 and ≤ 80 years 2. Subject or legal authorized representative is willing and able to give informed consent 3. Subject has a single targeted intracranial aneurysm that:

1. Is located in the internal carotid artery (ICA) distribution from petrous segment up to the terminus
2. Is able to be crossed with a standard 0.014" guide wire
3. Has unruptured saccular wide-neck (neck width ≥ 4 mm or dome-to-neck ratio < 2) or fusiform intracranial aneurysms size ≥10 mm
4. Has a vessel diameter ≥ 2.5 mm to ≤ 5.3 mm at both the proximal and distal segments where the implant will be placed 4. Subject is willing to comply with all scheduled follow-up visits and examinations per institutional standard of care

   Exclusion Criteria:

   Subject has a major surgery within previous 30 days or planned in the next 120 days after enrollment date 2. Previous intracranial implant associated with the symptomatic distribution within the past 12 weeks prior to treatment date 3. Subject has a non-target aneurysm treated within 30 days prior to study enrollment and a non-target aneurysm that requires treatment within 12 months.

   4. Subject has a planned treatment of a non-target aneurysm in the same vascular territory during participation in the study.

   5. Stenting, angioplasty, or endarterectomy of an extracranial (carotid or vertebral artery) or intracranial artery within 30 days prior to treatment date 6. Any previous coiling where it would interfere with the placement and proper apposition of the device 7. More than one intracranial aneurysm that requires treatment within 12 months 8. Contraindication to CT or MRI scans 9. Subject has severe neurological deficit (mRS score ≥ 3) that renders the subject incapable of living independently 10. Dementia or psychiatric problem that prevents the subject from completing required follow-up 11. Co-morbid conditions that may limit survival to less than 24 months 12. Other known serious concurrent medical conditions such as heart disease (e.g., atrial fibrillation/pacemaker, recent myocardial infarction, symptomatic congestive heart failure, and significant carotid artery disease), pulmonary disease, uncontrolled diabetes, progressive neurologic disorders, vasculitis, or subjects using immunosuppressants including corticosteroids.

   13. Female subjects who are pregnant or planning to become pregnant within the study period (all females of childbearing age must take a pregnancy test within 24 hours of treatment) and who are unwilling or unable to take adequate method of contraception for at least until the 12-month study follow-up*

   *If the subject becomes pregnant during her participation, the physician will have to evaluate the risk associated to her continuing participation to the rest of the study.

   14. Subject does not meet criteria or has any other contraindications listed in the DFU 15. Extra-cranial stenosis or parent vessel with stenosis >50% in the area proximal to the aneurysm 16. Subject with an intracranial mass (tumor, except meningioma, abscess, or other infection), or is undergoing radiation therapy for carcinoma or sarcoma of the head or neck region 17. Subject had a subarachnoid hemorrhage within 30 days prior to the enrollment date 18. Subject has a non-treated arterio-venous malformation (AVM) in the territory of the target aneurysm 19. Inability to understand the study or a history of non-compliance with medical advice 20. Current use of illicit substance 21. Enrollment in another trial involving an investigational product

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrolled, Not Treated (ENT) Population All subjects who sign the informed consent are considered enrolled and will be further screened by an angiogram to determine study eligibility.
  All subjects who are enrolled, have the pre-treatment angiogram, but never have the device enter their body, will be part of the Enrolled, Not Treated, angiogram (ENTa) population.
  For subjects that are enrolled, but exit the study before the pre-procedure angiogram, will be included in the Enrolled, Not Treated, no angiogram (ENTna) population. Members of the ENTna population will be followed to the time of study exit.
  Modified Intent to Treat Population The modified Intent to Treat (mITT) population will include all enrolled subjects for whom the Surpass Streamline FDS entered the body, regardless of deployment. The mITT subjects will be followed up to 5 years per protocol. Primary safety and efficacy analyses will be completed on the mITT population.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint. Percentage of subjects experiencing neurological death or major ipsilateral stroke in the treated vascular territory | 12 months
  Subjects experiencing neurological death or major ipsilateral stroke in the treated vascular territory through 12 months as adjudicated by an independent Clinical Events Committee (CEC).
Primary Efficacy Endpoint. Percentage of subjects with 100% occlusion (Raymond Class 1) without clinically significant stenosis defined as >50% stenosis of the parent artery | 12 months
  Subjects with 100% occlusion (Raymond Class 1) without clinically significant stenosis defined as >50% stenosis of the parent artery based on independent angiographic core laboratory evaluation of 12-month follow-up angiograms and having no retreatment of the target aneurysm through the 12 month follow-up visit timepoint.

SECONDARY OUTCOMES:
Secondary Safety Endpoints. Percent of subjects experiencing one or more SAEs | 60 months post-index procedure
  The secondary safety endpoint is the percent of subjects experiencing one or more SAEs through 60 months post-index procedure within the following categories (see definitions section of this protocol), as adjudicated by the Clinical Events Committee (CEC):
  * Device- and procedure-related SAEs at the peri-procedure timepoint and within 60 months of the index procedure as per visit schedule
  * Key neurological event of interest through 60 months post-procedure
Secondary Efficacy Endpoints. Surpass Streamline FDS technical success. The proportion of subjects in whom the Surpass Streamline implant(s) was delivered to cover the aneurysm neck. | Intraoperation
  All subjects who, at the end of their procedure, have the target aneurysm neck covered by the Surpass Streamline implant(s) will be considered technical successes. The percent and number of mITT subjects who are technical successes will be reported.
Secondary Efficacy Endpoints. Surpass Streamline FDS system success. The proportion of implants successfully delivered to the target location. | Intraoperation
  As part of the procedure case report form, investigators are asked if each used Surpass Streamline Flow Diverter was deployed to the target location. The percent and number of Surpass devices that enter a subject and are successfully deployed to the target location will be reported.
Secondary Efficacy Endpoints. Re-sheathing performance. The percent and number of Surpass devices that are successfully re-sheathed will be reported. | Intraoperation
  As part of the procedure case report form, investigators are asked if the Surpass Streamline Flow Diverter was re-sheathed successfully if the re-sheathing was applied. The percent and number of Surpass devices that are successfully re-sheathed will be reported.
Secondary Efficacy Endpoints. Functional status: change in the modified Rankin Scale (mRs) score compared to baseline. Percent of subjects who at follow-up exhibit improvement, worsening, or no change in their modified Rankin score compared to baseline. | 60 months
  Functional status: change in the modified Rankin Scale (mRs) score compared to baseline.
  The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 to 5. A separate category of 6 is usually added for patients who expire.
Secondary Efficacy Endpoints.Proportion of subjects with Raymond Class 1, 2 and 3 occlusions.The percent and number of mITT subjects in each Raymond class level at 12 and 36 months will be reported. | 12 and 36 months
  Proportion of subjects with Raymond Class 1, 2 and 3 occlusions.
  Raymond Classification will be determined on subtracted angiographic images as per clinical standard:
  * Raymond Class 1 = Complete Occlusion
  * Raymond Class 2 = Residual Neck
  * Raymond Class 3 = Residual Aneurysm.
Secondary Efficacy Endpoints. Incidence of retreatment through 60 months. The percent and number of mITT subjects who require retreatment, either with the Surpass Streamline Flow Diverter system or with another approach. | 60 months post-procedure
  Incidence of retreatment through 60 months
Secondary Efficacy Endpoints. The percent and number of mITT subjects who are recorded as having >50% stenosis of the parent artery at the target aneurysm location | 60 months
  Parent artery stenosis at the target aneurysm location >50%.
Secondary Efficacy Endpoints. The percent and number of mITT subject who are recorded as having >50% stenosis of their flow diverter | 60 months
  In-construct Surpass Streamline FDS stenosis >50%.
Secondary Efficacy Endpoints.The percent and number of mITT subject with any contrast opacification within the treated and previously fully occluded aneurysm on a subsequent angiographic study | 60 months post-procedure
  Target aneurysm recanalization

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Zhuhai People's Hospital, Zhuhai, Guangdong
  - The Second Affiliated Hospital of Guilin Medical College, Guilin, Guangxi
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Provincial People's Hospita, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Tangdu Hospital, Xi'an, Shaanxi
  - Xijing Hospital, Xi'an, Shaanxi
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong

IPD SHARING:
Plan to Share IPD: No
Terminated study with limited enrollments